CLINICAL TRIAL: NCT04285788
Title: Incidence and Outcomes Associated With the Management of Adenovirus Infections in Allogeneic Hematopoietic Cell Transplant Recipients: AdVance
Brief Title: Incidence and Outcomes Associated With the Management of Adenovirus Infections in Allogenic Hematopoietic Cell Transplant Recipients
Acronym: AdVance
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: AdVance
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Adenovirus Infections, Human
MeSH Terms: conditions — Adenovirus Infections, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To depict the incidence, outcomes and standards of care (SoC) of adenovirus (AdV) infections and associated practice patterns in allogeneic hematopoietic cell transplant recipients. It is expected that participating centers will be in the United Kingdom, France, Spain, Germany, and Italy.

ELIGIBILITY:
Inclusion Criteria:

* At least one AdV positive test, regardless of specimen within 6 months following the first allo-HCT
* Subjects first allo-HCT must have been performed between 1 January 2013 and 30 September 2015

Exclusion Criteria:

* AdV negative

Ages: 0 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: compromised of all allo-HCT recipients at participating centers during the pre-specified study period
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with non-relapse related mortality 3 and 6 months after first AdV Virema in paediatric allo-HCT recipients | 3 and 6 months after first adenovirus viremia
  To assess non-relapse related mortality 3 to 6 months after first adenovirus viremia.

SECONDARY OUTCOMES:
Number of participants who were hospitalized To assess the number of hospitalizations | 3 to 6 months
  To assess the number of hospitalizations, length of stay, and ICU stay.
The rate of adenovirus infection progression | 3 to 6 months
  To assess the rate of progression to disseminated adenovirus disease within the first year following allo-HCT